CLINICAL TRIAL: NCT03232619
Title: Safety and Efficacy Evaluation of CD19-CART Treatment for Refractory or Recurrent ALL
Brief Title: CD19-CART Treatment for ALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHBYCL001
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive CD19-CART cell immunotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CD19-CART with a murine scFv (Experimental): All enrolled patients in this arm will receive CD19-CART with a murine scFv.
  Interventions: Biological: CD19 CART
- humanized CD19-CART (Experimental): All enrolled patients in this arm will receive humanized CD19-CART.
  Interventions: Biological: CD19 CART

INTERVENTIONS:
Biological: CD19 CART — Patients will get one course of CART treatment with the dose of 0.5-5*10~6/KgBW.

SUMMARY:
This study aims to evaluate the safety and efficacy of a novel CD19-CART in the treatment of refractory or recurrent ALL.

DETAILED DESCRIPTION:
Chimeric antigen receptor T cell (CART) is a kind of engineered immunotherapy by transferring an artificial antigen binding receptor and also intercellular co-stimulating molecules into T cells. This kind of engineered T cells gains the ability to recognize antigen specific tumor cells and initiate the killing process in a HLA-independent way. CD19 is the specific cellular marker of B lineage acute leukemia (B-ALL), thus CD19-CART will be efficient in treating B lineage ALL. The investigators have constructed two kinds of CD19-CART. One is equipped with a murine CD19 scFv (single-chain variable fragmentt), while the other with a humanized scFv. This study aims to evaluate the safety and efficacy of both murine and humanized CD19-CART in treating refractory or recurrent ALL.

ELIGIBILITY:
Inclusion Criteria:

1. previously identified as CD19+ ALL.
2. ALL patients not eligible for allogeneic SCT or relapse after allogeneic SCT.
3. Expected survival >12W.
4. Creatinine < 2.5 mg/dl.
5. Alanine transaminase (ALT)/Aspartate Aminotransferase (AST) < 3x normal
6. Bilirubin <2.0 mg/dl
7. Voluntary informed consent is given.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Uncontrolled active infection.
3. Active hepatitis B or hepatitis C infection.
4. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
5. Previously treatment with any gene therapy products.
6. Any uncontrolled active medical disorder that would preclude participation as outlined.
7. HIV infection.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Radiological assessment | Month1 to Month12
  Radiological assessment of the therapeutic effect by systemic or local computed Tomography(CT) or positron emission tomography scan.

SECONDARY OUTCOMES:
The safety of CART immunotherapy | Day 1 to Week 4
  After CAR-T cell infusion,we will observe the potential adverse events, especially Cytokine Release Syndrome (CRS) and neurotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Yunxiao Xu, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Shanghai Bioray Inc., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No